CLINICAL TRIAL: NCT00762281
Title: A Prospective, Randomized, Multicenter Trial To Evaluate The Safety And Effectiveness Of The MEL 80 Excimer Laser Using LASIK (Laser In Situ Keratomileusis) For The Correction Of ≤ +6.0 D Of Hyperopia With Or Without Astigmatism Of +0.50 D To +3.50 D And MRSE ≤ +6.50 D
Brief Title: Safety and Effectiveness Study of the MEL 80 Excimer Laser Using LASIK in the Treatment of Hyperopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEL 80-2004-2
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Hyperopia
Keywords: Hyperopia; Laser In Situ Keratomileusis; Laser Therapy; Laser Corneal Surgery; Refractive Surgical Procedures; Ophthalmologic Surgical Procedure; Operative Surgical Procedures; Therapeutics
MeSH Terms: conditions — Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment of Hyperopic LASIK (Other): Treatment of Hyperopic corrections ≤ +6.0 D with or without Astigmatism of +0.50 to +3.50 D and MRSE ≤ +6.50 D.
  Interventions: Device: MEL 80 Hyperopic LASIK Treatment

INTERVENTIONS:
Device: MEL 80 Hyperopic LASIK Treatment — Treatment of Hyperopic corrections ≤ +6.0 D with or without Astigmatism of +0.50 to +3.50 D and MRSE ≤ +6.50 D.

SUMMARY:
The purpose of this study is to determine whether the MEL 80 Excimer Laser is effective in the treatment of hyperopia, when used as part of the Laser In Situ Keratomileusis (LASIK) procedure.

DETAILED DESCRIPTION:
LASIK has become one of the most common refractive eye procedures performed in the country. In the hyperopia procedure, a steepening occurs on the corneal surface, rather than the flattening procedure (myopic treatment). The surgeon will produce a standard keratomileusis flap using a microkeratome, exposing the corneal stroma. Recontouring under the flap is then accomplished by the removal of tissue from the stroma with the laser. This recontouring results in an altering of effective lens power of the central cornea, measured in diopters (D). The MEL 80 Excimer Laser System will be evaluated for its ability to create accurate and stable hyperopic refractive correction results.

ELIGIBILITY:
Inclusion Criteria:

* Naturally occurring hyperopia up to +6.0 D, with or without astigmatism of +0.50 D to +3.50 D at the spectacle plane, and MRSE ≤ +6.50 D;
* Have ≤ 0.75 D of latent hyperopia as determined by the difference between the preoperative MRSE and CRSE;
* A stable refraction for at least the last 12 months as documented by previous clinical records, i.e., the spherical and cylindrical portions of the manifest refraction have not progressed at a rate of more than 0.50 D during the year prior to the baseline examination in the eye to be treated;
* Hard contact lens wearers must have two central keratometry readings and two manifest refractions taken at least one week apart that do not differ by more than 0.50 D;
* Visual acuity correctable to at least 20/40 in both eyes;
* Operative eye must be targeted for emmetropia;
* At least 21 years of age;
* Willing and able to return for scheduled follow up examinations for 24 months after surgery;
* Sign and be given a copy of the written Informed Consent form.

Exclusion Criteria:

* A history of anterior segment pathology, including cataracts (in the operative eye);
* Severe dry eye syndrome unresolved by treatment;
* Residual, recurrent, active ocular or uncontrolled eyelid disease, corneal scars within the ablation zone or other corneal abnormality such as recurrent corneal erosion or severe basement membrane disease;
* Ophthalmoscopic signs of keratoconus (or keratoconus suspect);
* An ablation deeper than 250 microns from the corneal endothelium;
* Irregular or unstable (distorted/not clear) corneal mires on central keratometry readings;
* Blind in the fellow eye;
* Undergone previous intraocular or corneal surgery of any kind in the operative eye(s), including any type of excimer laser surgery for either refractive or therapeutic purposes;
* A history of ocular Herpes zoster or Herpes simplex keratitis;
* A history of steroid-responsive rise in intraocular pressure, glaucoma, or preoperative IOP >21 mm Hg;
* Diabetes, diagnosed autoimmune disease, connective tissue disease, or clinically significant atopic syndrome;
* Immunocompromised or use chronic systemic corticosteroid or other immunosuppressive therapy;
* Pregnant, lactating, or be of childbearing potential and not practicing a medically approved method of birth control;
* A known sensitivity to planned study medications;
* Participating in any other ophthalmic drug or device clinical trial during the time of this clinical investigation;
* At risk for angle closure or for developing strabismus postoperatively.
* For Fellow (Second) Eyes in Simultaneous Bilateral Treatment Procedures
* 1. Flap complications during the first eye's surgery such as a free cap, partial flap, thin flap, or irregular flap.
* 2. Epithelial defect exceeding 2 mm x 2 mm in dimension, or clinically significant debris in the interface between the flap and underlying stroma for the first eye.
* 3. Severe blepharospasm in the first eye that may have prevented or impeded the completion of the keratectomy and/or the laser ablation procedure.
* 4. Poor subject cooperation with instructions for the first eye's surgery and/or poor subject fixation on the laser fixation target.
* 5. Aborted LASIK procedure in the first eye or PRK was performed in the first eye because LASIK was not possible.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2004-07; Primary Completion 2006-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
At the point of stability, a minimum of 75% of eyes should have an achieved refraction within ± 1.00 D of the intended outcome, and at least 50% of eyes should be within ± 0.50 D of the intended outcome. | Point of stability
A minimum of 85% of eyes targeted for emmetropia should have an uncorrected visual acuity of 20/40 or better at the postoperative interval at which stability has been established. | Point of stability
A minimum of 95% of eyes should have a change of < 1.00 D in manifest refraction spherical equivalent (MRSE) between 2 refractions performed at least 3 months apart, and the mean rate of MRSE change per month should be < 0.04 D. | Point of stability
75% of eyes undergoing astigmatic treatment should be within ± 1.00 D of the attempted astigmatism correction by the point of stability. | Point of stability
Distance BSCVA of worse than 20/40 at the postoperative interval at which stability has been established should occur in less than 1.0% of eyes that had a BSCVA of 20/20 or better before surgery. | Point of stability
Loss of more than 2 lines of BSCVA should occur in less than 5.0% of eyes. | Point of stability
Less than 5% of eyes treated for sphere only should have a magnitude of postoperative manifest refractive astigmatism that varies from baseline cylinder by greater than 2.00 D at the postoperative interval at which stability has been established. | Point of stability
Incidence of Adverse Events to occur in less 1% of eyes | Postoperative visits

SECONDARY OUTCOMES:
Subject Satisfaction: As measured by a subjective questionnaire, and will be considered as a secondary efficacy variable. | Postoperative visits 3, 6, 9, 12, 18 and 24 months
Incidence of Complications | Postoperative visits
Patient Symptoms: As measured by a subjective questionnaire, will be considered as a secondary safety variable. | Preoperative and Postoperative visits 3, 6, 9, 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven Dell, MD, Principal Investigator — Texan Eye Care; John Doane, MD, Principal Investigator — Discover Vision Centers; Richard Hoffman, MD, Principal Investigator — Fine, Hoffman, and Packer LLC; Howard Fine, MD, Principal Investigator — Fine, Hoffman, and Packer LLC; Mark Packer, MD, Principal Investigator — FIne, Hoffman, and Packer LLC; David Tanzer, MD, Principal Investigator — US Navy Refractive Surgery Center, San Diego, CA; Steve Schallhorn, MD, Principal Investigator — US Navy Refractive Surgery Center, San Diego, CA; John Vukich, MD, Principal Investigator — Davis Duehr Dean Eye Clinic; Jon Dishler, MD, Principal Investigator — Dishler Laser Institute
Locations (6):
- United States (6):
  - US Navy Refractive Surgery Center, San Diego, California
  - Dishler Laser Institute, Greenwood Village, Colorado
  - Discover Vision Centers, Kansas City, Missouri
  - Fine, Hoffman, and Packer, Eugene, Oregon
  - Texan Eye Care, Austin, Texas
  - Davis Duehr Dean Eye Clinic, Madison, Wisconsin